CLINICAL TRIAL: NCT06099652
Title: A Multi-Centered, Randomized, Double-Blinded, Placebo-Controlled Phase II Clinical Trial, to Evaluate the Efficacy and Safety of 611 in Chinese Adults With Moderate to Severe Chronic Obstructive Pulmonary Disease.
Brief Title: Evaluation of 611 in Chinese Adults With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-611-COPD-II-01
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental): 611 300 mg Q2W, subcutaneous (SC) injection
  Interventions: Drug: 611 300 mg Q2W
- group B (Experimental): 611 450 mg Q2W, subcutaneous (SC) injection
  Interventions: Drug: 611 450 mg Q2W
- placebo group (Placebo Comparator): placebo Q2W, subcutaneous (SC) injection
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: 611 300 mg Q2W — 611 subcutaneous (SC) injection
  Arms: group A
Drug: 611 450 mg Q2W — 611 subcutaneous (SC) injection
  Arms: group B
Drug: Matching placebo — placebo subcutaneous (SC) injection
  Arms: placebo group

SUMMARY:
The primary objective of the study was to evaluate the efficacy and safety of 611 in Chinese adults with moderate to severe COPD.

DETAILED DESCRIPTION:
The maximum study duration was 28 weeks per participants, including a screening period of up to 4 weeks, a 16-week randomized treatment period, and a 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to understand and comply with the requirements of the study. and must participate voluntarily and sign the written informed consent.
2. Male or female adults ages 40 to 85 years old when signing the informed consent.
3. BMI≥16 kg/m2.
4. Documented diagnosis of COPD for at least one year prior to enrolment.
5. Post-bronchodilator FEV1/FVC < 0.70 and post-bronchodilator FEV1 % predicted >30% and ≤70%.
6. Current or former smokers with a smoking history of ≥10 pack-years or environmental exposure to biofuel fumes ≥10 years
7. Documented history of ≥ 2 moderate or ≥ 1 severe COPD exacerbations within 12 months prior to enrolment.
8. Background triple therapy (ICS + LABA + LAMA) for 3 months prior to randomization with a stable dose of medication for ≥1 month prior to randomization; Double therapy (LABA + LAMA) allowed if ICS is contraindicated.
9. Patients with blood eosinophils ≥200 cells/microliter at screening.
10. Female subjects of reproductive age (and their male partners) and male subjects (and their female partners) must use highly effective contraception throughout the study period and for at least 3 months after the last dose. The subjects had no plans to pregnancy, donate sperm or donate egg during the whole study period and for at least 3 months after the last dose.

Exclusion Criteria:

1. Significant pulmonary disease other than COPD (e.g., active tuberculosis，lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung disease, etc)
2. Diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
3. A current diagnosis of asthma or history of asthma according to the Global Initiative for Asthma (GINA) guidelines or other accepted guidelines.
4. Diagnosis of α-1 anti-trypsin deficiency.
5. Cor pulmonale, evidence of right cardiac failure
6. Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC).
7. A participant with a history of clinically significant renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, ophthalmologic, respiratory, gastrointestinal, cerebrovascular or other significant medical illness or disorder which, in the judgment of the Investigator, could interfere with the study or require treatment that might interfere with the study.
8. Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
9. Hypercapnia requiring Bi-level ventilation.
10. AECOPD as defined in inclusion criteria within 4 weeks prior to screening or randomization.
11. History of, or planned pneumonectomy or lung volume reduction surgery.
12. Treatment with oxygen of more than 12 hours per day.
13. Known with allergic or intolerant to mometasone furoate spray or 611/placebo.
14. Any reason which, in the opinion of investigator, would prevent the subject from participating in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pre-bronchodilator FEV1 at Week 16 | up to Week 16
  FEV1 is the Forced expiratory volume in one second at study site

SECONDARY OUTCOMES:
Change from baseline in Chronic Obstructive Pulmonary Disease assessment tool (CAT) score | up to Week 16
  Chronic Obstructive Pulmonary Disease assessment tool (CAT) score ranges from 0 to 40, a higher score indicating a higher impact on health status.
Change from baseline in St. George's Respiratory Questionnaire (SGRQ) total score | up to Week 16
  St. George's Respiratory Questionnaire (SGRQ) is a questionnaire designed to measure and quantify health-related health status in adult patients with chronic airflow limitation. A global score ranges from 0 to 100. Lower score indicates better quality of life.
Percentage of participants with a decrease in SGRQ total score of ≥ 4 points from baseline to Week 16 | up to Week 16
  St. George's Respiratory Questionnaire (SGRQ) is a questionnaire designed to measure and quantify health-related health status in adult patients with chronic airflow limitation. A global score ranges from 0 to 100. Lower score indicates better quality of life.
Annualized rate of moderate to severe COPD exacerbations in participants | up to Week 16
  Moderate or severe COPD exacerbation is defined by symptomatic worsening of COPD.
  Moderate：Use of systemic corticosteroids; and/or use of antibiotics; Severe：An inpatient hospitalization due to COPD
Time to first Moderate or severe COPD exacerbation | up to Week 16
  Moderate or severe COPD exacerbation is defined by symptomatic worsening of COPD.
  Moderate：Use of systemic corticosteroids; and/or use of antibiotics; Severe：An inpatient hospitalization due to COPD
Adverse events (AEs), measurement of vital signs，physical examination，electrocardiogram and laboratory tests at each visit. | Up to 24 Weeks
  The incidence and severity of treatment emergent adverse event (TEAE), including Serious Adverse Event (SAE), as well as clinical symptoms, and any abnormalities of vital signs, physical examinations，electrocardiogram，laboratory tests and, etc.
611 Concentration in Serum | Up to 24 Weeks
  The concentration of 611 in Serum
Percentage of Participants with Anti-drug Antibodies and Neutralizing Antibodies | Up to 24 Weeks
  Immunogenicity assessment will be based on Anti-drug Antibodies (ADAs) response and development of Neutralizing Antibodies (NABs). Percentage is calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-drug antibodies / number of evaluable participants * 100%.
Change in serum concentrations of PD variables | Up to 24 Weeks
  PD variables included Pulmonary and activation-regulated chemokine (PARC)，IgE，blood eosinophil counts and fibrinogen

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No